CLINICAL TRIAL: NCT03552978
Title: Tech and Telephone Smoking Cessation Treatment for Young Veterans With PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Tobacco Related Disease Research Program (Other); San Francisco Veterans Affairs Medical Center (U.S. Federal Agency); Northern California Institute of Research and Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-22551; NCI-2022-09681 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP)); 22634 (Other: University of California, San Francisco)
Record Dates: First submitted 2018-05-29; First posted 2018-06-12 (Actual); Results first posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tech-facilitated IC intervention (Experimental): After completing an initial 2-hour screening visit that includes a series of questionnaires assessing eligibility criteria and meeting with the study physician to review medical history, participants will be offered nicotine replacement therapy (NRT) at baseline (Week 0), per VA prescribing guidelines, nicotine dependence levels, and participant preference. Participants will then receive 8 counseling sessions (video or telephone). The first session lasts 45-60 min, and the remaining 7 sessions last 20-30 min. Participants will be asked to use the Stay Quit Coach (SQC) app between sessions, and the iCO® Smokerlyzer®
  Interventions: Behavioral: Tech-Facilitated IC Intervention
- VA Quitline (Active Comparator): After completing an initial 2-hour screening visit that includes a series of questionnaires assessing eligibility criteria and meeting with the study physician to review medical history, participants will be offered nicotine replacement therapy (NRT) at baseline (Week 0), per VA prescribing guidelines, nicotine dependence levels, and participant preference. Participants will also receive weekly proactive telephone sessions through the VA Quitline, a standard of care, proactive telephone quitline available to all veterans for up to eight weeks. Participants will initiate the first call and subsequent calls will be made by the Quitline counselor.
  Interventions: Behavioral: VA Quitline

INTERVENTIONS:
Behavioral: Tech-Facilitated IC Intervention — The Integrated Care (IC) treatment protocol for smoking cessation is a PTSD-informed intervention that has been adapted to be delivered over video or telephone and to incorporate technological components, including the Stay Quit Coach (SQC) smart phone application (app) which is a public domain, no-cost mobile app designed to complement the IC protocol with evidence-based tools to support smoking cessation. and the coVita Bedfont® Scientific Ltd iCO® Smokerlyzer® device and app which is a mobile carbon monoxide (CO) monitor that provides CO readings in order to self-monitor progress in quitting. The coVita mobile app is compatible with iOS &Android and used with the iCO® Smokerlyzer® to display CO readings. Content of sessions is consistent with that delivered in the IC treatment protocol for veteran smokers with post-traumatic stress disorder (PTSD).
  Arms: Tech-facilitated IC intervention
Behavioral: VA Quitline — The SFVAMC's standard of care referral service, known as the VA Quitline which involves weekly telephone sessions through the VA's proactive telephone Quitline, available to all veterans for up to 8 weeks.
  Arms: VA Quitline

SUMMARY:
This project aims to enhance the scalability of an office-based smoking cessation treatment protocol for veterans with PTSD, integrated care (IC), by adapting it to be delivered over the telephone and to incorporate mobile technology components. Mobile technology components include: (1) the Stay Quit Coach (SQC) mobile application (app), and (2) the iCO® mobile Smokerlyzer®, a smart phone-compatible carbon monoxide monitor.

DETAILED DESCRIPTION:
Eighty U.S. military veteran smokers with PTSD, ages 18-45, will be randomized to receive either: (1) the telephone-and technology-facilitated intervention (n=40), or (2) the current standard of care (referral to the VA telephone Quitline) (n=40) as a control. All participants will receive a baseline (Week 0) office visit and will optionally be prescribed nicotine replacement therapy (NRT). Participants in the intervention condition will receive eight 20- to 30-minute video or telephone counseling sessions and be asked to use the SQC app and iCO® Mobile Smokerlyzer®. Control participants will receive up to eight weekly proactive telephone sessions through the VA telephone Quitline. Assessments will occur at baseline (Week 0), treatment end (Week 8), and at three months (Week 12) and six months (Week 24) post-randomization. The primary aims of this pilot randomized controlled trial are: (1) to assess the feasibility and acceptability of the intervention; and (2) to assess the impact of the adapted IC intervention on treatment retention compared to treatment as usual (i.e., VA Quitline).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female veterans eligible for VA services
2. Ages 18 to 45 (inclusive)
3. Meets lifetime criteria for PTSD using the The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V)
4. Smoked at least 5 cigarettes per day for 15 of the past 30 days
5. Interested in smoking cessation and willing to receive interventions
6. A smartphone (iOS or Android) user and comfortable using a smartphone
7. Females must have a negative urine pregnancy test and must be practicing an effective method of birth control (e.g., surgically sterile, spermicide with barrier, male partner sterilization; or abstinent and agrees to continue abstinence or to use an acceptable method of contraception, as listed above, should sexual activity commence)
8. Ability to attend screening appointment in-person or via V-tel at San Francisco Veteran's Medical Center (SFVAMC) or an associated clinic and participate in 8 weekly sessions, follow-up sessions at Weeks 12 and 24, and monthly nicotine replacement check-ins

Modified inclusion criteria for remote screenings during Coronavirus Disease 2019 (COVID-19) pandemic:

7. Female participants will be required to provide a negative urine pregnancy test if they do not have a verified and reliable form of birth control (at the discretion of the PI). Pregnancy tests will be mailed to the participant and they will be asked to take a photo of the completed test and send it through an encrypted e-mail back to the study team in order to determine eligibility. Participants may also choose to complete urine pregnancy testing at VA lab. This will occur after verbal consent is given.

8. No longer required to be able to attend in-person screening appointment as everything will be done remotely. Potential recruits will need the ability to participate in telephone or secure, 2-way video conferencing "visits" for: Consent and Screening (Week 0), 8 weekly sessions, follow-up sessions at Weeks 12 and 24, and monthly nicotine replacement check-ins.

Exclusion Criteria:

1. Current, unstable psychotic or bipolar disorders
2. Dementia
3. Current, severe substance use disorder (SUD) deemed to be unstable by the study physician; individuals with SUD are eligible if their SUD is assessed to be in partial or full remission for 30 days or more at the time of screening, as assessed by Mini International Neuropsychiatric Interview (MINI) , chart review, and the principal investigator (PI).
4. Other psychiatric disorders judged to be unstable in the clinical judgment of the PI or study physician
5. Clinically significant unstable medical conditions, in the clinical judgment of the PI or study physician.
6. Female participants who are pregnant, intend to become pregnant during the study period, and/or are not using an effective method of birth control.
7. Concurrent participation in another smoking cessation study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Herbst, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco VA Medical Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Tech-facilitated IC Intervention: After completing an initial 2-hour screening visit that includes a series of questionnaires assessing eligibility criteria and meeting with the study physician to review medical history, participants will be offered nicotine replacement therapy (NRT) at Week 0, per VA prescribing guidelines, nicotine dependence levels, and participant preference. Participants will then receive 8 counseling sessions (telehealth). The first session lasts 45-60 min, and the remaining 7 sessions last 20-30 min. Participants will be asked to use the Stay Quit Coach (SQC) app between sessions, and the iCO® Smokerlyzer®
  Tech-Facilitated IC Intervention: The Integrated Care (IC) treatment protocol for smoking cessation is a PTSD-informed intervention that has been adapted to be delivered over video or telephone and to incorporate technological components, including the Stay Quit Coach (SQC) smart phone application which is a public domain, no-cost mobile app designed to complement the IC protocol with evidence-based tools to support smoking cessation. and the coVita Bedfont® Scientific Ltd iCO® Smokerlyzer® device and app which is a mobile carbon monoxide (CO) monitor that provides CO readings in order to self-monitor progress in quitting. The coVita mobile app is compatible with iOS &Android and used with the iCO® Smokerlyzer® to display CO readings. Content of sessions is consistent with that delivered in the IC treatment protocol for veteran smokers with post-traumatic stress disorder.
Period: Overall Study
Arm/Group | Tech-facilitated IC Intervention | VA Quitline
Started | 33 | 32
Completed | 30 | 31
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tech-facilitated IC Intervention | VA Quitline | Total
Number analyzed (Participants) | 33 | 32 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.27 (6.07) | 34.69 (4.95) | 33.97 (5.55)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 30 | 27 | 57
  Transgender Female | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 2 | 10
  Not Hispanic or Latino | 24 | 29 | 53
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 4 | 6 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 23 | 21 | 44
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 4 | 0 | 4
Sexual Orientation [Count of Participants; unit: Participants]
  Bisexual | 2 | 3 | 5
  Gay / Lesbian | 1 | 2 | 3
  Other | 0 | 1 | 1
  Straight / Heterosexual | 30 | 26 | 56

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Attending All Intervention Sessions
Description: Number of participants attending all intervention sessions.
Time Frame: over 8-week intervention period; calculated at Week 8 (post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Tech-facilitated IC Intervention | VA Quitline
Number analyzed (Participants) | 33 | 32
Participants | 18 | 3
Statistical Analysis 1: Comparison: Tech-facilitated IC Intervention vs VA Quitline; Test type: Superiority; p < .001, t-test, 2 sided; df - 63; Odds Ratio (OR) = 11.60

2. Primary Outcome: The Difference in Total Number of Treatment Sessions Attended Between the Experimental Treatment Condition and the Control Condition
Description: The difference in total number of treatment sessions attended between the experimental treatment condition and the control condition. Higher adherence rates suggest greater study/intervention feasibility and acceptability, and a large difference score would indicate greater feasibility/acceptability of one study condition over the other.
Time Frame: over 8-week intervention period; calculated at Week 8 (post-treatment)
Measure: Mean (Standard Deviation); unit: Sessions
Arm/Group | Tech-facilitated IC Intervention | VA Quitline
Number analyzed (Participants) | 33 | 32
Sessions | 6.18 (2.43) | 2.61 (2.69)
Statistical Analysis 1: Comparison: Tech-facilitated IC Intervention vs VA Quitline; Test type: Superiority; p < .001, t-test, 2 sided; df = 59; Mean Difference (Final Values) = 3.57

3. Primary Outcome: Acceptability Questionnaire
Description: Participants (in the intervention condition only) will complete a questionnaire developed by the investigators to rate the intervention protocol from 1-10 in terms of perceived helpfulness, understandability, and likelihood of use. The mean score (i.e., average of item ratings) will be reported for the participants in the intervention condition. Higher scores represent greater acceptability.
Time Frame: Week 8
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Tech-facilitated IC Intervention
Number analyzed (Participants) | 19
score on a scale | 8.67 (1.70)

4. Primary Outcome: Median Scores on the System Usability Scale (SUS)
Description: The SUS is a brief, reliable and valid instrument to measure perceptions of usability of technology devices. Items are rated on a scale from 0-5. An SUS total score is calculated by summing item ratings, and then multiplied the sum by 2.5. The maximum score on the SUS is 100, with higher scores reflecting greater usability. The SUS will be administered to the intervention condition only. Mean usability score will be reported.
Time Frame: Week 8
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Tech-facilitated IC Intervention
Number analyzed (Participants) | 19
score on a scale | 67.5 (19.47)

5. Primary Outcome: Median Scores on the Client Satisfaction Questionnaire-8 (CSQ-8)
Description: The CSQ-8 is an eight-item instrument designed to measure satisfaction with an clinical intervention. Items are rated on a scale from 1-4 and summed to for an CSQ-8 total score. Scores range from 8-32, with higher scores indicating greater satisfaction. The CSQ-8 will be administered to the intervention condition only. Mean satisfaction score will be reported.
Time Frame: Week 8 (post-treatment)
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Tech-facilitated IC Intervention
Number analyzed (Participants) | 19
score on a scale | 30 (4.5)

6. Secondary Outcome: Average Number of Cigarettes Smoked in the Past 30 Days at Weeks 0, 8, 12 and 24
Description: Self-reported use of cigarettes will be assessed with Timeline Follow-Back (TLFB) (past 30 days), which uses a calendar with specific anchor dates to identify the quantity and frequency of use. This outcome variable will be reported as the difference in cigarette use between the experimental treatment condition and the control condition.
Time Frame: Weeks 0, 8, 12, and 24
Population: Number analyzed at each session varies because not all participants attended all sessions.
Measure: Mean (Standard Deviation); unit: Cigarettes smoked in the past 30 days
Arm/Group | Tech-facilitated IC Intervention | VA Quitline
Number analyzed (Participants) | 33 | 32
Cigarettes smoked in the past 30 days
  Week 0 | 313.15 (178.22) | 353.97 (216.07)
  Week 8: number analyzed (Participants) | 20 | 21
  Week 8 | 210.76 (240.94) | 242.20 (254.70)
  Week 12: number analyzed (Participants) | 29 | 26
  Week 12 | 130.72 (150.74) | 253.96 (233.09)
  Week 24: number analyzed (Participants) | 28 | 29
  Week 24 | 131.25 (166.47) | 231.03 (236.48)
Statistical Analysis 1: Comparison: Tech-facilitated IC Intervention vs VA Quitline; We examined total Cigarettes smoked in the past 30 days using linear mixed models to account for non-independence (longitudinal data) and missing data. The null hypothesis was that the time by treatment group interaction would equal zero, indicating no difference in the change in cigarette use over time by treatment group; Test type: Superiority; p = .39, Mixed Models Analysis; df = 3, 152.11; Mean Difference (Final Values) = 90.28

7. Secondary Outcome: Timeline Follow-Back (TLFB): E-cigarettes
Description: Self-reported use of e-cigarettes will be assessed with TLFB (past 30 days), which uses a calendar with specific anchor dates to identify the quantity and frequency of use. This outcome variable will be reported as the difference in e-cigarette use between the experimental treatment condition and the control condition.
Time Frame: Weeks 0, 8, 12, and 24
Population: The number analyzed varies because not all participants attended all sessions.
Measure: Mean (Standard Deviation); unit: Days of e-cigarette use in the past 30
Arm/Group | Tech-facilitated IC Intervention | VA Quitline
Number analyzed (Participants) | 33 | 32
Days of e-cigarette use in the past 30
  Week 0 | 4.58 (10.08) | 2.97 (7.99)
  Week 8: number analyzed (Participants) | 17 | 13
  Week 8 | 0.88 (3.39) | 0 (0)
  Week 12: number analyzed (Participants) | 29 | 26
  Week 12 | 4.66 (9.90) | 3.58 (8.90)
  Week 24: number analyzed (Participants) | 28 | 29
  Week 24 | 3.82 (8.83) | 3.31 (8.25)
Statistical Analysis 1: Comparison: Tech-facilitated IC Intervention vs VA Quitline; We examined days of e-cigarette use in the previous 30 days using linear mixed models to account for non-independence (longitudinal data) and missing data. The null hypothesis was that the time by treatment group interaction would equal zero, indicating no difference in the change in e-cigarette use over time by treatment group; Test type: Superiority; p = .91, Mixed Models Analysis; df = 3, 140.87; Mean Difference (Final Values) = 0.49

8. Secondary Outcome: Timeline Follow-Back (TLFB): Chewing Tobacco
Description: Self-reported use of chewing tobacco will be assessed with TLFB (past 30 days), which uses a calendar with specific anchor dates to identify the quantity and frequency of use. This outcome variable will be reported as the difference in chewing tobacco use between the experimental treatment condition and the control condition.
Time Frame: Weeks 0, 8, 12, and 24
Population: The number analyzed varies because not all participants attended all sessions.
Measure: Mean (Standard Deviation); unit: Days of chewing tobacco use
Arm/Group | Tech-facilitated IC Intervention | VA Quitline
Number analyzed (Participants) | 33 | 32
Days of chewing tobacco use
  Week 0 | 0.48 (2.78) | 0 (0)
  Week 8: number analyzed (Participants) | 17 | 13
  Week 8 | 0 (0) | 0 (0)
  Week 12: number analyzed (Participants) | 29 | 26
  Week 12 | 0 (0) | 0 (0)
  Week 24: number analyzed (Participants) | 28 | 29
  Week 24 | 0.18 (0.94) | 0 (0)
Statistical Analysis 1: Comparison: Tech-facilitated IC Intervention vs VA Quitline; We examined days of chewing tobacco use in the previous 30 days using linear mixed models to account for non-independence (longitudinal data) and missing data. The null hypothesis was that the time by treatment group interaction would equal zero, indicating no difference in the change in chewing tobacco use over time by treatment group; Test type: Superiority; p = .66, Mixed Models Analysis; df = 3,199; Mean Difference (Final Values) = -0.18

9. Secondary Outcome: Change in Scores on the Fagerström Test for Nicotine Dependence (FTND)
Description: The FTND is a validated, 6-item self-report instrument that evaluates the intensity of physical addiction to nicotine. Three items are rated yes/no (0/1), and the other three items are rated on a scale from 0-3. Items are summed to yield a total score of 0-10, with higher scores reflecting greater nicotine dependence. This outcome variable will be reported as the difference in FTND total score between the experimental treatment condition and the control condition.
Time Frame: Weeks 0, 8, 12, and 24
Population: The number analyzed varies because not all participants attended all sessions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tech-facilitated IC Intervention | VA Quitline
Number analyzed (Participants) | 33 | 32
score on a scale
  Week 0 | 4.18 (2.30) | 4.66 (1.72)
  Week 8: number analyzed (Participants) | 18 | 28
  Week 8 | 2.67 (1.68) | 3.43 (2.25)
  Week 12: number analyzed (Participants) | 17 | 12
  Week 12 | 2.59 (1.42) | 2.08 (2.31)
  Week 24: number analyzed (Participants) | 13 | 12
  Week 24 | 2.92 (2.22) | 3.00 (2.09)
Statistical Analysis 1: Comparison: Tech-facilitated IC Intervention vs VA Quitline; We examined nicotine dependence using linear mixed models to account for non-independence (longitudinal data) and missing data. The null hypothesis was that the time by treatment group interaction would equal zero, indicating no difference in the change in nicotine dependence over time by treatment group; Test type: Superiority; p = .76, Mixed Models Analysis; df = 3, 102.04; Mean Difference (Final Values) = 0.33

10. Secondary Outcome: Biochemically Verified Point Prevalent Abstinence: 7-day
Description: Seven-day point prevalence abstinence rates will be confirmed by salivary cotinine levels. This outcome variable will be reported as the difference in abstinence rates between the experimental treatment condition and the control condition
Time Frame: Weeks 12 and 24
Population: The number analyzed varies because not all participants attended all sessions.
Measure: Count of Participants; unit: Participants
Arm/Group | Tech-facilitated IC Intervention | VA Quitline
Number analyzed (Participants) | 33 | 32
Participants
  Week 12: number analyzed (Participants) | 28 | 26
  Week 12 | 9 | 5
  Week 24: number analyzed (Participants) | 27 | 28
  Week 24 | 9 | 5
Statistical Analysis 1: Comparison: Tech-facilitated IC Intervention vs VA Quitline; Test type: Superiority; p = .28, Chi-squared — Week 12; df = 1; Odds Ratio (OR) = 1.99
Statistical Analysis 2: Comparison: Tech-facilitated IC Intervention vs VA Quitline; Test type: Superiority; p = .19, Chi-squared — Week 24; df = 1; Odds Ratio (OR) = 2.3

11. Secondary Outcome: Biochemically Verified Point Prevalence Abstinence: 30-day
Description: 30-day point prevalence abstinence rates will be confirmed by salivary cotinine levels. This outcome variable will be reported as the difference in abstinence rates between the experimental treatment condition and the control condition
Time Frame: Weeks 12 and 24
Population: The number analyzed varies because not all participants attended all sessions.
Measure: Count of Participants; unit: Participants
Arm/Group | Tech-facilitated IC Intervention | VA Quitline
Number analyzed (Participants) | 33 | 32
Participants
  Week 12: number analyzed (Participants) | 28 | 26
  Week 12 | 8 | 5
  Week 24: number analyzed (Participants) | 27 | 28
  Week 24 | 8 | 4
Statistical Analysis 1: Comparison: Tech-facilitated IC Intervention vs VA Quitline; Week 12; Test type: Superiority; p = .42, Chi-squared; df = 1; Odds Ratio (OR) = 1.68
Statistical Analysis 2: Comparison: Tech-facilitated IC Intervention vs VA Quitline; Week 24; Test type: Superiority; p = .17, Chi-squared; df = 1; Odds Ratio (OR) = 2.52

12. Secondary Outcome: Change in Scores on the PTSD Checklist for DSM 5 (PCL-5)
Description: The PCL-5 is a 20-item self-report measure that assesses the severity of the twenty DSM-V symptoms of PTSD. Items are rated on a 1-5 scale and summed to compute a total score, with higher scores representing greater severity of PTSD symptoms. The total score can range from 0 to 80. This outcome variable will be reported as the difference in PCL-5 total score between the experimental treatment condition and the control condition.
Time Frame: Weeks 0, 8, 12, and 24
Population: The number analyzed varies because not all participants attended all sessions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tech-facilitated IC Intervention | VA Quitline
Number analyzed (Participants) | 33 | 32
score on a scale
  Week 0 | 35.94 (17.29) | 37.38 (20.53)
  Week 8: number analyzed (Participants) | 18 | 28
  Week 8 | 40.17 (17.66) | 33.00 (20.31)
  Week 12: number analyzed (Participants) | 17 | 12
  Week 12 | 38.12 (21.27) | 26.08 (19.42)
  Week 24: number analyzed (Participants) | 13 | 12
  Week 24 | 29.08 (18.52) | 25.42 (15.50)
Statistical Analysis 1: Comparison: Tech-facilitated IC Intervention vs VA Quitline; We examined days of changes in PTSD symptoms using linear mixed models to account for non-independence (longitudinal data) and missing data. The null hypothesis was that the time by treatment group interaction would equal zero, indicating no difference in the change in PTSD symptoms over time by treatment group; Test type: Superiority; p = .58, Mixed Models Analysis; df = 3, 100.51; Mean Difference (Final Values) = 3.66

13. Other Pre Specified Outcome: Timeline Follow-Back (TLFB): Other Tobacco Products
Description: Self-reported use of any other tobacco products will be assessed with TLFB (past 30 days), which uses a calendar with specific anchor dates to identify the quantity and frequency of use. This outcome variable will be reported as the difference in use of other tobacco products between the experimental treatment condition and the control condition.
Time Frame: Weeks 0, 8, 12, and 24
Population: Unfortunately there was a miscommunication between the study plan and the questionnaire and "Other tobacco use" was not collected. This was not a pre-specified secondary outcome measure per protocol, rather an exploratory measure.
Arm/Group | Tech-facilitated IC Intervention | VA Quitline
Number analyzed (Participants) | 0 | 0

14. Other Pre Specified Outcome: Proportion of Participants Recruited Based on Region
Description: The difference in recruitment rates among residents of rural versus urban areas. Higher recruitment rates suggest greater study and intervention feasibility, and a large difference score would indicate greater feasibility based on type of residential area.
Time Frame: over 8-week intervention period; calculated at Week 8 (post-treatment)
Population: Participant census tract was not collected, so this measure cannot be reported. This was not a pre-specified primary outcome measure per protocol, and was originally an an exploratory measure.
Arm/Group | Tech-facilitated IC Intervention | VA Quitline
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 Weeks
Description: There were no adverse events to report in this study.
Groups:
- Tech-facilitated IC Intervention: After completing an initial 2-hour screening visit that includes a series of questionnaires assessing eligibility criteria and meeting with the study physician to review medical history, participants will be offered nicotine replacement therapy (NRT) at Week 0, per VA prescribing guidelines, nicotine dependence levels, and participant preference. Participants will then receive 8 counseling sessions (telehealth). The first session lasts 45-60 min, and the remaining 7 sessions last 20-30 min. Participants will be asked to use the Stay Quit Coach (SQC) app between sessions, and the iCO® Smokerlyzer®
  Tech-Facilitated IC Intervention: The Integrated Care (IC) treatment protocol for smoking cessation is a PTSD-informed intervention that has been adapted to be delivered over video or telephone and to incorporate technological components, including the Stay Quit Coach (SQC) smart phone application which is a public domain, no-cost mobile app designed to complement the IC protocol with evidence-based tools to support smoking cessation. and the coVita Bedfont® Scientific Ltd iCO® Smokerlyzer® device and app which is a mobile carbon monoxide (CO) monitor that provides CO readings in order to self-monitor progress in quitting. The coVita mobile app is compatible with iOS &Android and used with the iCO® Smokerlyzer® to display CO readings. Content of sessions is consistent with that delivered in the IC treatment protocol for veteran smokers with post-traumatic stress disorder (PTSD).
Arm/Group | Tech-facilitated IC Intervention | VA Quitline
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/32
Other Adverse Events (participants affected / at risk) | 0/33 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-18): https://cdn.clinicaltrials.gov/large-docs/78/NCT03552978/Prot_SAP_000.pdf
  • Informed Consent Form (2019-08-20): https://cdn.clinicaltrials.gov/large-docs/78/NCT03552978/ICF_001.pdf